CLINICAL TRIAL: NCT05276765
Title: Peri-implant Soft Tissue Conditioning of Immediate Posterior Implants by CAD/CAM Socket Sealing Abutments (A Randomized Controlled Clinical Trial)
Brief Title: Peri-implant Soft Tissue Conditioning of Immediate Posterior Implants by CAD/CAM Socket Sealing Abutments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elgendi, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11122
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Implant Site Reaction
Keywords: immediate posterior implants, socket sealing abutments

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM customized Socket Sealing Abutment (Experimental): Anatomically formed healing abutments that can solve many of the problems inherent to immediate posterior implant placement and to optimize the conditioning of supra implant tissue architecture enhancing the emergence profile of the final implant restoration
  Interventions: Procedure: cad/cam socket sealing abutment
- Standard healing abutment (Active Comparator): Standard healing abutment will be inserted after removal of cover screw after immediate implant insertion and then a muco-periosteal flap will be reflected for the primary closure of the socket and sutured around the standard healing abutment.
  Interventions: Procedure: standard healing abutment

INTERVENTIONS:
Procedure: cad/cam socket sealing abutment — Anatomically formed healing abutments that can solve many of the problems inherent to immediate posterior implant placement and to optimize the conditioning of supra implant tissue architecture enhancing the emergence profile of the final implant restoration
  Arms: CAD/CAM customized Socket Sealing Abutment
Procedure: standard healing abutment — Standard healing abutment will be inserted after removal of cover screw after immediate implant insertion and then a muco-periosteal flap will be reflected for the primary closure of the socket and sutured around the standard healing abutment.
  Arms: Standard healing abutment

SUMMARY:
One of the major challenges one clinician can face while performing immediate placement on posterior area, is the ability of obtaining a hermetic primary closure of the soft tissue. The use of socket sealing abutment may provide advantages in maintaining the existing soft tissue architecture, preserving crestal bone height and reducing the risk of premature loading of the immediate implant during healing

DETAILED DESCRIPTION:
One of the major challenges one clinician can face while performing immediate placement on posterior area, is the ability of obtaining a hermetic primary closure of the soft tissue. This technical skill is nearly always combined with invasive surgical procedures and significant post op recovery (displacement of the muco-gingival line, periosteal releasing incision, flaps, sutures, membrane stabilization, …).the use of customized healing abutment may provide advantages in maintaining the existing soft tissue architecture, preserving crestal bone height and reducing the risk of premature loading of the immediate implant during healing.

Moreover, customized healing abutment can passively accommodate the definitive prosthesis with minimal or no pressure placement preventing biological or mechanical trauma during the prosthetic phases. This may lead to better long-term tissue stability and avoid the pain perceived by the patients from compression of tissues in case of standard healing abutment.

the primary aim of this randomized controlled clinical study is to clinically evaluate and compare the soft tissue outcomes of final immediate implant restorations placed in maxillary posterior sites that were conditioned by CAD/CAM fabricated socket sealing abutments versus standard healing abutments.

The secondary aim of this study is to radiographically assess peri-implant bone level changes of the final immediate implant restorations placed in maxillary posterior sites for the two experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patients ≥18 years old. 2. Non-restorable maxillary posterior teeth with intact adjacent teeth. 3. Sufficient bone to insert a dental implant with a minimum length of 8 mm and at least 3.5 mm in diameter.

  4. Type1 extraction socket according to Elian et al, 200742 (Labial bone plate and associated soft tissues are completely intact).

  5. Sufficient mesio-distal, bucco-lingual, and inter-occlusal space for placement of the definite restoration.

  6. Adequate oral hygiene (full mouth plaque score < 25% and full mouth bleeding score < 25%).

  7. Patients capable of understanding and giving informed consent.

Exclusion Criteria:

* 1. Alcohol or drug abusers. 2. Heavy smokers (> 10 cigarettes/day). 3. Presence of acute periapical infections. 4. Radiotherapy to the head and neck region for malignancy. 5. Bruxism or TMJ dysfunction. 6. Intake of drugs affecting bone metabolism. 7. Uncontrolled diabetic patients. 8. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Pink esthetic score | one year of follow up
  clinical evaluation of soft tissue profile around the implant restorations with minimum score of 0 and maximum score of 10

SECONDARY OUTCOMES:
Functional implant prosthodontic score | one year of follow up
  clinical evaluation of implant restoration assembly and radiographic crestal bone loss with minimum score of 0 and maximum score of 10

CONTACTS AND LOCATIONS:
Overall Officials: Amina Zaki, PhD degree, Principal Investigator — Professor in Fixed Prosthodontics department, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elgendi MM, Hamdy ISE, Sallam HI. Peri-implant soft tissue conditioning of immediate posterior implants by CAD-CAM socket sealing abutments: a randomized clinical trial. BMC Oral Health. 2025 Jan 17;25(1):83. doi: 10.1186/s12903-024-05417-w. PMID 39819325